CLINICAL TRIAL: NCT05686798
Title: Phase I Study of Replication-Competent Adenovirus-Mediated Double Suicide Gene Therapy With Stereotactic Radiosurgery in Patients With Recurrent or Progressive High Grade Astrocytomas
Brief Title: Adenovirus Mediated Suicide Gene Therapy With Radiotherapy in Progressive Astrocytoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Tobias Walbert, MD, PhD, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HFHS-21-02
Record Dates: First submitted 2022-11-16; First posted 2023-01-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Malignant Glioma of Brain; Astrocytoma; Malignant Astrocytoma; Brain Tumor; Glioma; Brain Cancer; Glioblastoma; Glioblastoma Multiforme; GBM
MeSH Terms: conditions — Astrocytoma; Brain Neoplasms; Glioma; Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ad5-yCD/mutTKSR39rep-ADP adenovirus and fSRS Arm (Experimental): Subjects will receive a single intratumoral injection of the Ad5-yCD/mutTKSR39rep-ADP adenovirus at one of three dose levels beginning at 1 x 1011 vp and escalating in half-log (3-fold) increments to 1 x 1012 vp, along with the same dose of fractionated stereotactic radiosurgery until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Biological: Ad5-yCD/mutTKSR39rep-ADP adenovirus and fractionated stereotactic radiosurgery (fSRS)

INTERVENTIONS:
Biological: Ad5-yCD/mutTKSR39rep-ADP adenovirus and fractionated stereotactic radiosurgery (fSRS) — Ad5-yCD/mutTKSR39rep-ADP adenovirus will be injected intratumoral

SUMMARY:
The primary goal of this Phase I study is to determine the maximum tolerated dose of oncolytic adenovirus mediated double suicide-gene therapy in combination with fractionated stereotactic radiosurgery in patients with recurrent high-grade astrocytoma undergoing resection.

DETAILED DESCRIPTION:
Detailed study description:

Patients with recurrent glioblastoma (GBM) or progressive high grade astrocytoma who are scheduled to undergo repeat surgery are eligible. After the removal of as much tumor tissue as possible, a modified oncolytic adenovirus is injected into the wall of the resection cavity and any residual tumor tissue. The goal of this study is to determine the maximum tolerated dose (MTD) of the injected adenovirus. This treatment is combined with a combination of oral 5-fluorocytosine (5-FC) and valganciclovir (vGCV) prodrug therapy. Following the surgery, patients will be treated with fractionated radiosurgery (fSRS). Patients will be monitored for 30 days before they start on next line anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with radiologic evidence of intracranial recurrence or progression of a previously diagnosed high-grade astrocytoma.

   To be eligible for this trial, the subjects must have:
   * Histologically documented glioblastomas or anaplastic astrocytoma prior to the debulking surgery that is suspicious to have progressed on imaging. An interval of at least 3 months must have elapsed since the completion of the most recent course of radiation while at least 4 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen.
   * Patients must be ≥ 18 years of age, able to provide informed consent and express a willingness to meet all the expected requirements of the protocol for the duration of the study.
   * Must have recovered from toxicity (grade 2 or less) of prior therapy.
   * Eligible for partial or total resection of the recurrent tumor
   * No anticipated physical connection between post-resection tumor cavity and cerebral ventricle
   * Karnofsky performance status (KPS) ≥ 60 at time of surgery
   * No prior treatment of the tumor with gene or virus therapy, immunotherapy, brachytherapy, or implants of polymers containing chemotherapeutic agents (e.g. Gliadel Wafer)
   * No immunosuppressive or immune disorder
   * Baseline organ function testing intact
   * Patients who are candidates for surgical debulking (re-resection) following recurrence of diseases based on multidisciplinary evaluation by neurosurgeons, radiation oncologists, neuro-radiologists, and neuro-oncologists.
2. Subjects must have adequate baseline organ function, as assessed by the following laboratory values, within 30 days before initiating the study therapy:

   * Adequate renal function with creatinine clearance ≥ 50 mL/min/m2
   * Platelet count ≥ 100,000/μL
   * Absolute neutrophil count ≥ 1,000/μL
   * Hemoglobin > 10.0 g/dL
   * Bilirubin < 1.5 mg/dL; SGOT and SGPT < 2.5 times upper limit of normal (ULN).
3. Women of child-bearing potential will be required to practice birth control for the duration of the treatment and for at least 90 days after surgery with intratumor virus inoculation. Men must use barrier protection for the duration of treatment and for at least 90 days after surgery with intratumor virus inoculation treatment.

Exclusion Criteria:

* Acute infection. Acute infection is defined by any viral, bacterial, or fungal infection that has required active treatment and caused oral temperature >38.5oC and/or clinically significant leukocytosis
* Serum antibodies to human immunodeficiency virus (HIV)
* Previous history of liver disease including autoimmune or viral hepatitis
* Positive serologic test for Hepatitis B or C at baseline
* Immunosuppressive therapy except for corticosteroid use
* Serious medical or psychiatric illness or concomitant medication, which, in the judgment of the investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial
* Impaired immunity or susceptibility to serious viral infections
* Pregnant or lactating females
* Allergy to any product used on the protocol
* Patient is not able to undergo a brain MRI.
* Patients who are not eligible for debulking surgery or resection of recurrent disease will be considered ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 30 days
  The primary objective is to determine the maximum tolerated dose of injected of Ad5-yCD/mutTKSR39rep-ADP adenovirus into the resection cavity at the time of surgery.

SECONDARY OUTCOMES:
1. Assessment of antitumor immune response | Pre-surgery (day 0), 3, 7, 14, 21, 30, 90 days.
  Assessment of antitumor immune response by serum levels of interferon-gamma (IFN-γ) measured by ELISA and will be described by pico-gram per milliliter (pg/mL).
2. Assessment of change in antitumor immune response by peripheral blood monoclonal cell (PBMC) counts | Pre-surgery (day 0), 3, 7, 14, 21, 30, 90 days.
  Assessment of change in antitumor immune response by peripheral blood monoclonal cell (PBMC) counts measured by flow cytometry
Assessment of antitumor immune response by using antibodies against surface markers | Pre-surgery (day 0), 3, 7, 14, 21, 30, 90 days.
  Assessment of antitumor immune response by using antibodies against surface markers (CD3, CD56, CD4, CD8, CD45, CD69).

OTHER OUTCOMES:
Quality of life as assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 | Pre-surgery (day 0), 30 days, 90 days
  Assessment of quality of life (QOL) by using the European Organization for Research and Treatment of Cancer (EORTC) tools consisting of the EORTC QLQ-C30
Quality of life as assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-BN20 | Pre-surgery (day 0), 30 days, 90 days
  Assessment of quality of life (QOL) by using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-BN20

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Walbert, MD, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ene CI, Fueyo J, Lang FF. Delta-24 adenoviral therapy for glioblastoma: evolution from the bench to bedside and future considerations. Neurosurg Focus. 2021 Feb;50(2):E6. doi: 10.3171/2020.11.FOCUS20853. PMID 33524949
- [Background] Mitchell LA, Lopez Espinoza F, Mendoza D, Kato Y, Inagaki A, Hiraoka K, Kasahara N, Gruber HE, Jolly DJ, Robbins JM. Toca 511 gene transfer and treatment with the prodrug, 5-fluorocytosine, promotes durable antitumor immunity in a mouse glioma model. Neuro Oncol. 2017 Jul 1;19(7):930-939. doi: 10.1093/neuonc/nox037. PMID 28387849
- [Background] Kiyokawa J, Wakimoto H. Preclinical And Clinical Development Of Oncolytic Adenovirus For The Treatment Of Malignant Glioma. Oncolytic Virother. 2019 Oct 24;8:27-37. doi: 10.2147/OV.S196403. eCollection 2019. PMID 31750274
- [Background] Oldfield EH, Ram Z, Culver KW, Blaese RM, DeVroom HL, Anderson WF. Gene therapy for the treatment of brain tumors using intra-tumoral transduction with the thymidine kinase gene and intravenous ganciclovir. Hum Gene Ther. 1993 Feb;4(1):39-69. doi: 10.1089/hum.1993.4.1-39. PMID 8384892
- [Background] Chen SH, Shine HD, Goodman JC, Grossman RG, Woo SL. Gene therapy for brain tumors: regression of experimental gliomas by adenovirus-mediated gene transfer in vivo. Proc Natl Acad Sci U S A. 1994 Apr 12;91(8):3054-7. doi: 10.1073/pnas.91.8.3054. PMID 8159705
- [Background] Freytag SO, Rogulski KR, Paielli DL, Gilbert JD, Kim JH. A novel three-pronged approach to kill cancer cells selectively: concomitant viral, double suicide gene, and radiotherapy. Hum Gene Ther. 1998 Jun 10;9(9):1323-33. doi: 10.1089/hum.1998.9.9-1323. PMID 9650617